CLINICAL TRIAL: NCT02160366
Title: Profile Related Evidence to Determine Individualized Cancer Therapy (PREDICT) Program in Advanced Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: LAB10-0441; 3UL1RR024148-04S1 (NIH)
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Molecular profiling; Biomarker data; Data analysis; Tumor marker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected may include blood, fresh tumor tissue, urine, saliva, bone marrow, pleural fluid, ascites, skin or hair follicle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biomarker/Molecular Data Collection and Analyzation: Advanced cancer participants
  Interventions: Other: Biomarker Research

INTERVENTIONS:
Other: Biomarker Research — Research studies on new biomarkers conducted on previously banked blood and/or tumor tissue. Samples collected may include blood, fresh tumor tissue, urine, saliva, bone marrow, pleural fluid, ascites, skin or hair follicle.

SUMMARY:
The goal of this laboratory research study is to collect and analyze treatment, molecular profiling and biomarker data. The results of the data analysis will be used to better understand how to characterize tumors and identify therapies that may be tailored to individual patients and to identify and/or predict side effects that may occur and/or predict which therapies may be best for participants. Research may also be done on your existing tissue to identify new biomarkers.

DETAILED DESCRIPTION:
Molecular Profiling/Deep Sequencing:

Molecular profiling is the classification of tissue based on the expression of certain genes within a tumor that might predict how the tumor responds to therapy. Deep sequencing is a more detailed type of molecular profile that allows for a more focused analysis of individual genes.

Biomarker Data:

A characteristic that is measured and evaluated as an indicator of normal biologic processes, disease processes or pharmacologic responses to a therapeutic intervention.

Study Participation:

If you agree to take part in this study, information from your medical record will be collected. The information that researchers will collect includes your medical history, chemotherapy schedule(s), as well as the results of any tests, procedures, and/or therapies you may have had. Your responses to the therapies, your side effects, and the results of any diagnostic tests performed during therapy will also be collected.

Researchers want to learn if they could have better predicted your response to therapy using the information collected in this study and/or better predict side effects from your treatment.

The data collected from your medical record will be stored in a password-protected database at MD Anderson to be used in research related to this study for up to 10 years.

In addition, research studies on new biomarkers may be conducted on your previously banked blood and/or tumor tissue. Samples collected may include blood, fresh tumor tissue, urine, saliva, bone marrow, pleural fluid, ascites, skin or hair follicle.

Your name, medical record number, and any other personal identifiable information collected from your medical record will be replaced with a code number. No identifying information will be directly linked to the data collected from your medical record. Only the doctor who is in charge of this study, and select members of their research staff, will have access to the code numbers and be able to link any of the data back to you.

Use of Samples:

Before your banked tissue samples can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of MD Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at MD Anderson, including research involving your tissue samples from this bank, must first be approved by the IRB.

Your tissue samples will be given a code number. No identifying information will be directly linked to your samples. Only the researcher in charge of the bank will have access to the code numbers and be able to link the samples to you. This is to allow medical data related to the samples to be updated as needed. Other researchers using your samples will not be able to link this data to you.

Length of Study:

Your participation in this study will be over after either the data, blood, tumor tissue samples, and/or archived tumor samples are analyzed.

This is an investigational study.

Up to 2000 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred to the Clinical Center for Targeted Therapy are potentially eligible for recruitment.

Exclusion Criteria:

n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the Clinical Center for Targeted Therapy at UT MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-09-27 (Actual); Primary Completion 2020-09-27 (Estimated); Study Completion 2020-09-27 (Estimated)

PRIMARY OUTCOMES:
Comparison of Biomarker Profiling to Treatment Outcome | 2 months
  For correlating marker profiles with response to treatment, univariate and multivariate (multiple covariates) logistic regression used, with response status taken as outcome variable. Distributions of time-to-event outcomes estimated using Kaplan-Meier curves, and these distributions compared among groups using log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Weitz J, Nishizaki D, Liau J, Patel J, Ng I, Sun S, Ramms D, Zou J, Wishart B, Rull J, Baumgartner J, Kelly K, White R, Veerapong J, Hosseini M, Patel H, Botta G, Gutkind JS, Tiriac H, Kato S, Lowy AM. Cyclin-Dependent Kinase 4/6 Inhibition as a Novel Therapy for Peritoneal Mucinous Carcinomatosis With GNAS Mutations. J Clin Oncol. 2025 Feb 20;43(6):705-715. doi: 10.1200/JCO.24.00511. Epub 2024 Oct 16. PMID 39413348
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org